CLINICAL TRIAL: NCT02726672
Title: Fatigue and Inspiratory Muscles Training Against Resistance in Patients With Multiple Sclerosis With Severe Disabilities
Brief Title: Fatigue and Inspiratory Muscles Training in Patients With Multiple Sclerosis
Acronym: AIRSEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC-P0043; 2015-A01451-48 (Other: ANSM)
Record Dates: First submitted 2016-03-22; First posted 2016-04-04 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Multiple Sclerosis
Keywords: inspiratory muscles; multiple sclerosis; rehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Respiratory rehabilitation (Experimental): Respiratory rehabilitation: Powerbreathe training of the inspiratory muscles at home twice a day (2 sessions of 30 inspirations / day) during 10 weeks
  Interventions: Device: respiratory rehabilitation using Powerbreathe
- control group (No Intervention): No respiratory rehabilitation

INTERVENTIONS:
Device: respiratory rehabilitation using Powerbreathe — 10 minutes 2 times a day : 30 inspirations per session during 10 weeks
  Arms: Respiratory rehabilitation

SUMMARY:
The purpose of this study is to assess the effect of a training of the inspiratory muscles against resistance at home during 10 weeks in multiple sclerosis patients with a severe disability.

DETAILED DESCRIPTION:
Patients will be informed about the study procedures during a follow-up consultation or an hospitalization in a Physical and Rehabilitation Medicine Unit. If they give their informed consent to participate in the study, an investigator will randomize them into one of the 2 arms of the study. This study consists of 3 visits. The first visit (inclusion) is planned at day 0, the second visit 10 weeks later and the third 3 months after day 0. A patient who is randomized in the experimental arm will have to follow 10 weeks of rehabilitation of the inspiratory muscles at home between first and second visit. During this period, investigators will call these patients once a week to assess the compliance with the rehabilitation. The patients who have been randomized in the control group will not follow this rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Patient with remitting or progressive multiple sclerosis defined by McDonald criteria revised in 2005, with an EDSS between 6 and 7,5
* Aged between 18 and 65 years
* Patients able to maintain the Powerbreathe
* Not to have had a flare-up since at least 6 weeks
* Patients at least 4 weeks since a corticoid bolus
* Patients at least 6 weeks since a botulinum toxin injection
* Patients at least 4 weeks since a pulmonary infection
* Questionnaire EMIF-SEP >= 55
* Patients given their informed consent
* Patients who benefit or are affiliated to a social security regimen

Exclusion Criteria:

* Patients with neurologic antecedents other that multiple sclerosis
* Patients with respiratory disorders other than those induced by multiple sclerosis
* Patients with orthopedic, cardiac, and rheumatologic invalidating antecedents
* Patients with comprehension or cognitive disorders impeding the realization of rehabilitation
* Pregnant women
* Patients under legal guardianship, or safeguard of justice
* Patients participating or planning participate within the 3 months of the study to another clinical research project

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Fatigue graded according to EMIF-SEP questionnaire | 3 months
  EMIF-SEP questionnaire (French valid version of the Fatigue Impact Scale, self-administered questionnaire to measure fatigue in multiple sclerosis patients)

SECONDARY OUTCOMES:
Sleep disorders graded according to the Epworth Sleepiness Scale | 3 months
Quality of life graded according to the SEP-59 questionnaire | 3 months
  SEP-59 questionnaire (french validated self-administered questionnaire to assess quality of life in multiple sclerosis patients)
Maximal inspiratory pressure graded according to the Black and Hyatt method | 3 months
  respiratory manometer according to Black and Hyatt method
Maximal expiratory pressure graded according to Black and Hyatt method | 3 months
  respiratory manometer according to Black and Hyatt method
Forced vital capacity (FVC) graded with a portable spirometer | 3 months
Tidal volume graded with a portable spirometer | 3 months
Forced expiratory volume in one second (FEV1) graded with a portable spirometer | 3 months
FEV1/ FVC ratio graded with a portable spirometer | 3 months
Energy consumption during repeated effort | 3 months
  Metamax 3B
Depression graded according to the French version of the Beck Depression Inventory Fast-Screen | 3 months
  French version of the Beck Depression Inventory Fast-Screen, validated scale in multiple sclerosis
Swallowing problems graded according to the DYMUS score | 3 months
Level of disability graded by the EDSS (Expanded Disability Status Scale) | 3 months
  These functional parameters will enable the assessment of the level of disability by a clinical examination
Collection of the drug treatments received evaluated by a questionnaire | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Donzé, MD, Principal Investigator — Hospital Group of the Catholic Institute of Lille
Locations (1):
- Hospital Group of the Catholic Institute of Lille, Lomme, France

IPD SHARING:
Plan to Share IPD: No